CLINICAL TRIAL: NCT06483243
Title: A Randomized, Open-label, Single Oral Dosing, Two-sequence, and Two-period Crossover Study to Evaluate the Pharmacokinetics and Safety Between the Administration of CKD-383 and the Co-administration of CKD-501, D745, and D150 for Healthy Subjects in Fed State
Brief Title: Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic of CKD-501, D745, and D150 for Healthy Subjects in Fed State.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A101_05BE2315
Record Dates: First submitted 2024-06-13; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): * Phase 1: CKD-501 1 tablet, D745 1 tablet, D150 2 tablets(Reference)
  * Phase 2: CKD-383 2 tablets(Test)
  Interventions: Drug: Test: CKD-383, Reference1: Duvie Tab. 0.5mg, Reference2: Jardiance tablets 25 mg, Reference3: GLUCOPHAGE XR TAB. 1000MG
- Group B (Experimental): * Phase 1: CKD-383 2 tablets(Test)
  * Phase 2: CKD-501 1 tablet, D745 1 tablet, D150 2 tablets(Reference)
  Interventions: Drug: Test: CKD-383, Reference1: Duvie Tab. 0.5mg, Reference2: Jardiance tablets 25 mg, Reference3: GLUCOPHAGE XR TAB. 1000MG

INTERVENTIONS:
Drug: Test: CKD-383, Reference1: Duvie Tab. 0.5mg, Reference2: Jardiance tablets 25 mg, Reference3: GLUCOPHAGE XR TAB. 1000MG — At around 8 a.m., take Test drug or Reference drug 1,2,3(oral) with 200 mL of water at room temperature.
  Other Names: Test: CKD-383, Reference1: CKD-501, Reference2: D745, Reference3: D150

SUMMARY:
This is a Randomized, open-label, single oral dosing, two-sequence, and two-period crossover study to evaluate the pharmacokinetics and safety between the administration of CKD-383 and the co-administration of CKD-501, D745, and D150 for healthy subjects in fed state

DETAILED DESCRIPTION:
Participants were randomly assigned in a 1:1 ratio. The patients are prescribed oral administration of the appropriate IP(2 or 4 tablets in single dose: actual medication)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 65 years
* Based on screening, no congenital or chronic disease, who have no athological symptoms or findings(If necessary, EEG, ECG, chest and gastroscopy or gastrointestinal radiation, Examination)
* within 5 years prior to the start of the trial(Period 1 administration) of any clinically significant mental medical history
* Other inclusion criteria, as defined in the protocol

Exclusion Criteria:

* who has taken drug metabolism enzyme induction and inhibitory drugs, such as barbitale drugs, within 30 days prior to the start of the trial (Period 1 administration)
* Other exclusive criteria, as defined in the protocol

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
AUCt of Lobeglitazone, Empagliflozin, Metformin | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization
Cmax of Lobeglitazone, Empagliflozin, Metformin | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization

SECONDARY OUTCOMES:
AUC∞ of Lobeglitazone, Empagliflozin, Metformin | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization
Tmax of Lobeglitazone, Empagliflozin, Metformin | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization
T1/2 of Lobeglitazone, Empagliflozin, Metformin | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization
CL/F of Lobeglitazone, Empagliflozin, Metformin | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization
Vd/F of Lobeglitazone, Empagliflozin, Metformin | 0 hour ~ 48 hour after drug administration
  Pharmacokinetic characterization

CONTACTS AND LOCATIONS:
Overall Officials: Yun Hwan Oh, PI, Principal Investigator — Chung-Ang University Gwangmyeong Hospital
Locations (1):
- Chung-Ang University Gwangmyeong Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No